CLINICAL TRIAL: NCT02495610
Title: A Prospective Single-centre Trial Investigating Novel Parameters for the Prediction of Ventriculoperitoneal Shunting Efficacy in Patients With Idiopathic Normal Pressure Hydrocephalus
Brief Title: Novel Parameters for the Prediction of Ventriculoperitoneal Shunting Efficacy in Patients With iNPH
Acronym: iNPH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-Nr. 2014-0423
Record Dates: First submitted 2015-06-23; First posted 2015-07-13 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: NPH; Gait analysis; neuropsychology; micturition diary; MRI
MeSH Terms: interventions — Gait Analysis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gait analysis and MRI (Other): * Gait analysis: Intervention: Treadmill with pressure sensors (FDM-THM-M-System (Force distribution method-treadmill); 'Zebris' medical GmbH), study-specific, but routine procedures.
  * MRI: Intervention: Performed in a scanner at the University Hospital with standard MRI compatibility procedures; study specific is only the additional MRI after the CSF release with spinal tap or drainage.
  Interventions: Other: Gait analysis and MRI:

INTERVENTIONS:
Other: Gait analysis and MRI: — * Gait analysis: Treadmill with pressure sensors (FDM-THM-M-System; 'Zebris' medical GmbH), study-specific, but routine procedures.
  * MRI: Performed in a scanner at the University Hospital with standard MRI compatibility procedures; study specific is only the additional MRI after the CSF release with spinal tap or drainage.

SUMMARY:
INPH is a chronic, progressive disease characterised by enlarged ventricles in the absence of elevated intracranial pressure. Patients often present with the Hakim triad comprising gait disturbance, dementia and urinary incontinence. Treatment consists of ventriculoperitoneal (VP) shunting reducing the cerebrospinal fluid (CSF) volume in the central nervous system (CNS); a generally safe and well tolerated procedure nevertheless invasive in nature and associated with surgical risk. The currently used diagnostic algorithms to predict surgery outcome by testing patients before and after a diagnostic spinal tap temporarily reducing the CSF volume in the CNS are of wide variability and limited validity. Developing measures to accurately diagnose and select patients for intervention is thus of great importance. The objective of this study is to define and validate a diagnostic algorithm for the selection of patients with symptoms compatible with iNPH for shunt surgery.

DETAILED DESCRIPTION:
Idiopathic normal pressure hydrocephalus (iNPH) is an important differential diagnosis of dementia in the elderly patients. It is characterised by an enlargement of the ventricular system and can lead to cognitive deficits, gait disturbance and incontinence. Treatment consists of a ventriculoperitoneal shunt. A major challenge is the identification of patients who suffer from iNPH and who will benefit from shunt surgery. Typically, cerebrospinal fluid (CSF) is withdrawn by a spinal tap, and walking speed and steps per distance are measured before and thereafter. In patients who benefit from the test tap the diagnosis iNPH is made and the indication for shunt surgery is ascertained. The diagnostic procedure is not standardised.

Little is known about the examinations and time-points suited best to predict surgery outcome. Thus, patients may undergo surgery who do not benefit, and patients who would benefit may be missed.

This study aims at defining a diagnostic algorithm to improve the prediction of surgery outcome in patients supposed to suffer from iNPH. In 25 serial patients, motor function will be analysed in detail by functional tests and a treadmill-based analysis before and after the test tap at different time-points. In addition, neuropsychological tests and MRI investigations (DWI and pw) will be done, and patients will fill-out a micturition diary. Patients who do not respond to the test tap will be offered a lumbar drainage for continuous CSF release as diagnostic escalation with repeated tests thereafter. Patients who finally undergo shunt surgery will be re-assessed to identify those who responded to surgery. Thereby, post-hoc analyses will identify those parameter(s) that had the best predictive value for surgery outcome. To confirm the parameters derived from such exploratory analyses, these parameters will be validated in another series of 25 patients.

The results of this study have the potential to improve the clinical routine and to provide a strategic advantage for the University Hospital Zurich.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Age 50 years or above
* Impaired walking function for at least 3 months, onset at/ after 40 years of age.
* MRI or CT with enlarged ventricular system (Evans' index ≥0.30) without evidence of moderate or severe cortical atrophy.
* Eligible for shunt surgery.
* Eligible for analysis of gait, neuropsychological and urological function.
* Subjects must be able to understand the patient information sheet and comply with the requirements of the protocol.

Exclusion Criteria:

* Previous intracranial disorder or surgery.
* Contraindications to surgery or MRI
* Contraindications to the testing of gait, bladder or neuropsychological function.
* Presence of concomitant disease which might reasonably account for the clinical symptoms or radiological findings.
* Worsening of walking function secondary to any other condition occurring during the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-06; Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Gait Analysis on treadmill by foot print plate and overground walking by time keeping | 3 months
  a composite of the following measurements: Step width, step length, Foot rotation, double stance phase, cadence, velocity (Timed 25 Foot Walk, endurance (6 minute walking test)

SECONDARY OUTCOMES:
MRI | 3 months
  a composite of fractional anisotropy, mean diffusivity, parallel diffusivity, radial diffusivity
Urological function by micturition diary | 3 months
  a composite of the following informations: number of voiding, number of incontinence episodes, number of urgency episodes
Neuropsychology by validated testing | 3 months
  a composite of response inhibition and switching (stroop test), working memory (wechsler memory scale), verbal fluency (Regensburg word fluency), figural fluency (number of unique designs and repetitions of the same figure), divided and focused attention (TMT A, TMT B)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Prof., Principal Investigator — University of Zurich
Locations (1):
- University Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Hakim S, Adams RD. The special clinical problem of symptomatic hydrocephalus with normal cerebrospinal fluid pressure. Observations on cerebrospinal fluid hydrodynamics. J Neurol Sci. 1965 Jul-Aug;2(4):307-27. doi: 10.1016/0022-510x(65)90016-x. No abstract available. PMID 5889177
- [Background] Marmarou A, Young HF, Aygok GA, Sawauchi S, Tsuji O, Yamamoto T, Dunbar J. Diagnosis and management of idiopathic normal-pressure hydrocephalus: a prospective study in 151 patients. J Neurosurg. 2005 Jun;102(6):987-97. doi: 10.3171/jns.2005.102.6.0987. PMID 16028756
- [Background] Relkin N, Marmarou A, Klinge P, Bergsneider M, Black PM. Diagnosing idiopathic normal-pressure hydrocephalus. Neurosurgery. 2005 Sep;57(3 Suppl):S4-16; discussion ii-v. doi: 10.1227/01.neu.0000168185.29659.c5. PMID 16160425
- [Background] Stolze H, Kuhtz-Buschbeck JP, Drucke H, Johnk K, Diercks C, Palmie S, Mehdorn HM, Illert M, Deuschl G. Gait analysis in idiopathic normal pressure hydrocephalus--which parameters respond to the CSF tap test? Clin Neurophysiol. 2000 Sep;111(9):1678-86. doi: 10.1016/s1388-2457(00)00362-x. PMID 10964082